CLINICAL TRIAL: NCT04657770
Title: Telerehabilitation Early After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Moss Rehabilitation Research Institute (Other)
Responsible Party: Principal Investigator, Steven C. Cramer, MD, FAAN, FAHA, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-000994
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Results first posted 2023-04-12 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Stroke
Keywords: telerehab; telerehabilitation; telehealth; brain plasticity
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: All enrollees will receive telerehabilitation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Telerehabilitation (Experimental): Patients will receive 36 treatment sessions over 6 weeks, consisting of 3 sessions/week that are supervised rehab therapy sessions (which begin with a 30-minute videoconference with the licensed OT or PT), alternating with 3 sessions/week of unsupervised rehab therapy sessions whereby the patient follows the instructions on the screen to engage in rehab therapy. Because patients sometimes miss a session, e.g., due to a conflict, we allow up to 8 weeks for patients to complete their 36 rehab therapy sessions.
  Interventions: Device: Telerehabilitation

INTERVENTIONS:
Device: Telerehabilitation — The telerehabilitation system will deliver rehabilitation treatment sessions via a secured internet-connected computer. A major component of the system is the use of games to promote therapeutically relevant movements. The subject will perform daily assigned remote-based telerehabilitation games and exercises and 5 minutes of stroke education, all guided by the telerehabilitation system. During some of the sessions, therapists will initiate a videoconference with the subject's telerehabilitation system to discuss progress, issues, and revise treatment plans as needed.

SUMMARY:
The purpose of this research study is to assess the feasibility of initiating telerehab in early stages after stroke during patient admission to an inpatient rehabilitation facility. Patients will complete 36 sessions of telerehab 6 days/week up to 8 weeks with a telehealth system provided in their hospital room and at their home. The system will include rehabilitation activities/exercises, education, and assessments to evaluate the patient experience and measure patient outcomes at the end of a 6-week course of telerehab.

DETAILED DESCRIPTION:
Stroke is a major cause of disability. Loss of movement is a major part of this. Studies show that high doses of rehabilitation therapy can reduce disability, but many patients do not receive this, e.g., due to obstacles such as difficulty accessing care. The research team has previously found that telerehabilitation is an effective way to deliver care and improve outcomes. These prior studies were performed after hospital discharge, when patients were already back at home. The current study aims to extend this work by introducing telerehabilitation to the bedside of patients admitted to an inpatient rehabilitation facility. In this study, key areas of interest include issues related to, and the clinical effects of, telerehabilitation that is started during the rehab admission and is continued after discharge in the patient's home.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Stroke that has been radiologically verified
3. Arm motor FM score <56 (out of 66) at initial visit
4. Box & Block Test score with affected arm is at least 3 blocks in 60 seconds at initial visit
5. Informed consent and behavioral contract signed by the subject
6. Admitted to California Rehabilitation Institute or MossRehab for stroke rehabilitation

Exclusion Criteria:

1. A major, active, coexistent neurological or psychiatric disease (e.g., alcoholism or dementia)
2. A major medical disorder that substantially reduces the likelihood that a subject will be able to comply with all study procedures
3. Severe depression, as defined as Geriatric Depression Scale Score >10 at initial visit
4. Significant cognitive impairment, as defined as Montreal Cognitive Assessment score <22 (lower score permitted if due to aphasia with approval from Dr. Cramer)
5. Deficits in communication that interfere with reasonable study participation
6. Lacking visual acuity, with or without corrective lens, of 20/40 or better in at least one eye
7. Life expectancy <6 months
8. Pregnant
9. Receipt of Botox to arms, legs, or trunk in the preceding 6 months, or expectation that Botox will be administered to the arm, leg, or trunk within 3 months of study enrollment
10. Unable to successfully perform study procedures/therapy or attend study visits, or expectation of noncompliance with study procedures/therapy
11. Non-English speaking, such that subject does not speak sufficient English to comply with study procedures
12. Expectation that subject will not have a single domicile address during the 6 weeks of therapy that has either Verizon wireless reception or a home WiFi network and that has space for the telerehab system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - California Rehabilitation Institute, Los Angeles, California
  - Moss Rehabilitation Research Institute, Elkins Park, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
A deidentified dataset will be shared with appropriate personnel after the main study manuscript is published.
Supporting Information: Study Protocol, SAP
Time Frame: Likely starting 1-2 years after study completion, lasting for several years thereafter.
Access Criteria: Data will be shared using common data formats with appropriate personnel.

REFERENCES:
- [Derived] Edwards D, Kumar S, Brinkman L, Ferreira IC, Esquenazi A, Nguyen T, Su M, Stein S, May J, Hendrix A, Finley C, Howard E, Cramer SC. Telerehabilitation Initiated Early in Post-Stroke Recovery: A Feasibility Study. Neurorehabil Neural Repair. 2023 Feb-Mar;37(2-3):131-141. doi: 10.1177/15459683231159660. Epub 2023 Mar 6. PMID 36876946

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telerehabilitation
Started | 19
Completed | 15
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Completed training but withdrew before follow-up testing due to change in medical status | 1

BASELINE CHARACTERISTICS:
Arm/Group | Telerehabilitation
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Fugl-Meyer Arm Motor Score From Baseline to End of Treatment (60 Days)
Description: Measure of arm impairment. Scores range from 0-66, with higher numbers reflecting less arm impairment.
  We will be measuring change in scores from baseline to end of treatment (60 days).
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telerehabilitation
Number analyzed (Participants) | 15
units on a scale | 18.07 (10.85)

ADVERSE EVENTS:
Time Frame: For each subject, from baseline to 10 weeks post-enrollment
Arm/Group | Telerehabilitation
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 4/19
Other Adverse Events (participants affected / at risk) | 2/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telerehabilitation (N=19)
Sepsis (General disorders) | 1 (1) — Sepsis, not related to study procedures
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pneumonia, not related to study procedures
Recurrent stroke (Nervous system disorders) | 1 (1) — recurrent stroke, not related to study procedures
Shoulder injury (Musculoskeletal and connective tissue disorders) | 1 (1) — Rotator cuff injury sustained during home health therapy (therapist not part of study), unrelated to stud procedures
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telerehabilitation (N=19)
Nausea (Nervous system disorders) | 1 (1) — Nausea when wearing prism glasses during TR
Depression (Psychiatric disorders) | 1 (1) — Depressive symptoms when being asked questions related to depression during standardized testing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT04657770/Prot_SAP_002.pdf